CLINICAL TRIAL: NCT05966714
Title: Neonatal Electrical Activity at Different Altitude Levels: A Prospective Observational Cohort Study
Brief Title: Neonatal Electrical Activity at Different Altitude Levels
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: 20230509-z
Record Dates: First submitted 2023-06-14; First posted 2023-08-01 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Altitude Hypoxia; Neonatal Encephalopathy
Keywords: altitude; neonate; Amplitude integrated electroencephalography
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Lijiang(2500m)
  Interventions: Device: aEEG
- Group 2: Shangri-La (3500 m)
  Interventions: Device: aEEG

INTERVENTIONS:
Device: aEEG — amplitude-integrated electroencephalography

SUMMARY:
In this study, the objective is to compare neonatal cerebral electrical activity within 3 days after birth across different altitude areas using amplitude-integrated electroencephalography (aEEG), and establish reference value for each altitude level.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton term infants (gestational age between 37 0/7 and 41 6/7 weeks) born in the participating hospital.
2. Infants appear well as defined by normal vital signs (heart rate ranging from 110 to 180 beats/min, respiratory rate ranging from 30 to 60 breaths/min, temperature ranging from 36.5°C to 37.5°C), absence of signs of illness such as cyanosis, respiratory distress and heart murmur.
3. The mother is permanent residence of the current altitude level and live in the study area for the entire duration of pregnancy.

Exclusion Criteria:

1. Need for supplemental oxygen or assisted ventilation.
2. Any evidence of intrauterine distress such as meconium-stained amniotic fluid, Apgar score <7 at 1 or 5 min.
3. Referred to neonatal intensive care unit or neonatology department for any reason other than observation.
4. With major congenital anomaly.
5. Probes cannot be properly placed due to scalp lesions or hematomas.
6. Reject or withdraw from the study.

Ages: 0 Hours to 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy neonates at different altitude levels
Sampling Method: Probability Sample
Enrollment: 531 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
Differences in aEEG indicators in neonates within three days after birth at different altitudes | within three days after birth
  aEEG data are acquired by aEEG device. This minimum and maximum value is used as the preliminary smoothing value for that specific time point. Next, a three-order low-pass filter is employed to further refine the preliminary values, and a phase compensation algorithm is applied to restore temporal information and obtain smoothed boundaries.For further analyzing the aEEG data, a total of 63 signal features were extracted to reflect the spectral density aspects by the Auto-Neo-EEG pipeline.

SECONDARY OUTCOMES:
Establish reference values for each altitude level | within three days after birth
  If significant differences exist across altitude levels, the 3rd, 10th, 50th, 75th, 90th, and 97th percentile for upper and lower threshold of aEEG will be established for each group separately. Otherwise a combined reference interval will be provided using the average value of lower limit value.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Yangfang Li, Kunming, Yunnan
  - Children Hospital of Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No